CLINICAL TRIAL: NCT05597293
Title: Effect of Introduction of FreeStyle Libre Monitoring on Glycaemic Control in People with Type 2 Diabetes Mellitus (T2DM)
Brief Title: FreeStyle Libre Monitoring in T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hull (Other)
Responsible Party: Principal Investigator, Thozhukat Sathyapalan, Professor, University of Hull
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 301630
Record Dates: First submitted 2022-10-24; First posted 2022-10-28 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Type2diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- FreeStyle Libe 2 (Active Comparator): Participants in this group will wear the FreeStyle Libre 2 device
  Interventions: Device: Glucose monitoring using FreeStyle Libre 2
- FreeStyle Libre pro iQ (Active Comparator): Participants in this arm will wear the FreeStyle Libre pro iQ device
  Interventions: Device: Glucose monitoring using FreeStyle Libre pro iQ

INTERVENTIONS:
Device: Glucose monitoring using FreeStyle Libre 2 — Glucose monitoring in patients with type 2 diabetes using FreeStyle Libre 2
  Arms: FreeStyle Libe 2
Device: Glucose monitoring using FreeStyle Libre pro iQ — Glucose monitoring in patients with type 2 diabetes using FreeStyle Libre pro iQ
  Arms: FreeStyle Libre pro iQ

SUMMARY:
The goal of this clinical trial is to learn if blood sugar monitoring using a FreeStyle Libre device can improve overall Diabetes control in people with Type 2 Diabetes.

The main questions it aims to answer are:

* What is the effect of monitoring using the FreeStyle Libre device for a period of 12 weeks on the blood sugar control of people with Type 2 Diabetes?
* Can monitoring using the FreeStyle Libre device improve the quality of life of people with Type 2 diabetes?

Participants will be asked to wear one of two brands of FreeStyle Libre devices. In one group, participants will have 3 visits, while those in the second group, they will have 4 visits.

Researchers will compare the improvement in the sugar control for the individuals but also compare between the 2 groups.

DETAILED DESCRIPTION:
This is a prospective, randomised, open-labelled, non-CTIMP, pilot study. Participants meeting the inclusion criteria and who have consented to participate in the study will be randomised on a 1:1 ratio to receive either Libre 2 or Libre pro iQ. Randomisation will be carried out using an online randomisation tool to allocate a participant to a treatment group.

The study will consist of three visits (Libre 2 arm) and four visits (Libre pro iQ arm). The study will be completed over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females living with type 2 diabetes mellitus (T2DM) who are aged ≥ 18 and ≤ 75 years
* On one or more non-insulin glucose lowering agent(s)
* HbA1c ≥ 69 mmol/mol
* Able to provide written informed consent

Exclusion Criteria:

* Participants with a life expectancy of less than 1 year
* Participants with cognitive dysfunction or neurological disorder, which will interfere with regular, flash glucose monitoring
* Participants with chronic kidney disease (CKD) with eGFR < 45ml/min/1.73m2 or decompensated liver disease or decompensated congestive cardiac failure
* Myocardial infarction in the preceding 3 months or if percutaneous coronary intervention planned in the next 6 months
* Participants on supra-physiological doses of steroids, for example, Prednisolone for the treatment of Rheumatoid arthritis
* Participants on active dialysis or planned for dialysis treatment during the study
* Currently participating in another device or drug study that could affect glucose measurements or management
* Women who are pregnant, breastfeeding or planning to become pregnant. Women should use a reliable form of contraception throughout the study
* Participants who are already using continuous glucose monitoring (CGM)
* Participants who have pacemakers, implanted cardioverter defibrillator devices or neurostimulators
* Participants with an allergy to medical grade adhesive
* A blood transfusion in the preceding 3 months or a planned blood transfusion during the course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with a change in HbA1c of 5.5 mmol/mol or more | 12 weeks
  The number of participants with a change in HbA1c of 5.5 mmol/mol or more at the end of the study compared to baseline HbA1c

SECONDARY OUTCOMES:
Change in the Diabetes Quality of Life (DQOL) score | 12 weeks
  Change in Diabetes Quality of Life (DQOL) score from baseline to end of the study. The total scores range from 0 (lowest possible quality of life) to 100 (highest possible quality of life). Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, FRCP,FACP, Principal Investigator — University of Hull
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Academic diabetes, Endocrinology and metabolism, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies MJ, D'Alessio DA, Fradkin J, Kernan WN, Mathieu C, Mingrone G, Rossing P, Tsapas A, Wexler DJ, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2018. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2018 Dec;41(12):2669-2701. doi: 10.2337/dci18-0033. Epub 2018 Oct 4. PMID 30291106
- [Background] Deshmukh H, Wilmot EG, Gregory R, Barnes D, Narendran P, Saunders S, Furlong N, Kamaruddin S, Banatwalla R, Herring R, Kilvert A, Patmore J, Walton C, Ryder REJ, Sathyapalan T. Effect of Flash Glucose Monitoring on Glycemic Control, Hypoglycemia, Diabetes-Related Distress, and Resource Utilization in the Association of British Clinical Diabetologists (ABCD) Nationwide Audit. Diabetes Care. 2020 Sep;43(9):2153-2160. doi: 10.2337/dc20-0738. Epub 2020 Jul 15. PMID 32669277
- [Background] Edge J, Acerini C, Campbell F, Hamilton-Shield J, Moudiotis C, Rahman S, Randell T, Smith A, Trevelyan N. An alternative sensor-based method for glucose monitoring in children and young people with diabetes. Arch Dis Child. 2017 Jun;102(6):543-549. doi: 10.1136/archdischild-2016-311530. Epub 2017 Jan 30. PMID 28137708